CLINICAL TRIAL: NCT04732260
Title: Prenatal Treatment of Congenital Cytomegalovirus Infection With Letermovir Randomized Against Valaciclovir - STEP 1
Brief Title: Prenatal Treatment of Congenital Cytomegalovirus Infection With Letermovir Randomized Against Valaciclovir - CYMEVALIII STEP1
Acronym: CYMEVAL3-STEP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP180592; 2020-002924-35 (EudraCT Number)
Record Dates: First submitted 2021-01-24; First posted 2021-02-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2022-02

CONDITIONS: Pregnant Women Undergoing TOP; TOP - Failed Attempted Termination of Pregnancy
Keywords: Cytomegalovirus; Pregnant women
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- letermovir (Experimental): Maternal administration of 1 tablet of Letermovir (240 mg or 480 mg /day) during 3 days before TOP
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Each patient will receive 1 tablet of Letermovir (240 mg or 480 mg /day) during 3 days before TOP.
  5 women will receive 240 mg. 5 women will receive 480 mg.

SUMMARY:
In the model of the perfused cotyledon, Letermovir crosses the placenta to reach appropriate fetal concentration. The cotyledon model can only be performed in the third trimester placenta. Although it is probable that the transplacental passage in the second trimester is in the same range than the one found in the 2th trimester, it needs to be confirmed. The study will be divided in 2 steps: step 1 will study the Letermovir transplacental transfer in the second trimester and step 2 will test the efficacy of letermovir to inhibit replication in infected fetuses.

Main objective To measure the Letermovir transplacental transfer in the second trimester and its accumulation in the amniotic fluid and the placenta in the second trimester

Primary end point:

Concentrations reached in fetal blood relative to EC50 of letermovir.

DETAILED DESCRIPTION:
The eligible population of step 1 will be pregnant women in their second trimester of pregnancy and undergoing TOP for any fetal abnormality and no evidence of placental dysfunction.

Letermovir (LTM) is a new anti CMV drug, manufactured by Merck that:

* is highly efficient in vitro against CMV (more than ganciclovir the gold standard drug)
* is as efficient as valganciclovir to cure CMV infection and highly efficient as a prophylaxis to avoid CMV infection and disease in bone marrow transplated patients
* is very well tolerated
* has no data from the use in pregnant women and animal studies are insufficient with respect to fetotoxicity, but no specific concern in pregnant women arises from its safety profile
* crosses the placenta in the ex vivo model of the human perfused cotyledon to reach efficient fetal concentration

In this STEP 1 study, we elected to test 2 Letermovir dosages:

* 240 mg given orally once a day. Based on 10% rate of letermovir transplacental passage as demonstrated in the cotyledonon model, we calculated that the dosage of 240 mg given once a day to the pregnant woman should be suffisent to reach efficient concentration in fetal blood.
* 480 mg /day given orally once a day. 480 mg per day is the recommended dose to prevent CMV infection in bone marrow transplanted patients;

The risks added by the study are those of letermovir: nausea, diarrhea and vomiting (frequent), hypersensitivity, loss of appetite, headache, vertigo, abdominal pain, ALT and AST increase, muscule spasm, blood creatinine increase, fatigue, peripheral edema (very rare). The expected benefit for the women is: none.

Women and obstetrician investigator will sign the written consent for the trial.

* Validation of inclusion and non-inclusion criteria will be assessed by the obstetrician investigator as follows:
* age, weight, height and medical history will be collected.
* Inquiry on maternal concomitant treatment(s)
* Blood sampling: (4 ml altogether)
* 1 Heparinate Lithium tube (2 ml) for measurements of urea, creatinine, creatinine clearance, liver enzyme (ALAT ASAT GGT PAL), bilirubine
* 1 EDTA tube of 2 ml for full blood test count These measurements will be done in the biochemistry laboratory of the investigating site.

When validation of inclusion and non-inclusion criteria is done (all the criteria will be available on the day of the baseline visit), the woman receives the tablets of letermovir. They will be allocated either 240 mg or 480 mg up until termination of pregnancy. 5 women will receive 240 mg. In order to have variation in the time elapsed between administration and sampling, it will be asked to 3 women to take the drug every morning and to 2 patients to take the drug every evening. 5 women will receive 480 mg. This time, it will be asked to 2 women to take the drug every morning and to 3 patients to take the drug every evening.

Hence, the day of TOP, patients who take the drug every evening will have the largest delay between the last intake and blood sampling. The patients who take the drug every morning should take the last tablet early in the morning the day of TOP and latest 4 hours before the blood sampling.

After the baseline visit, there will be one other visit just before TOP; the obstetrician investigator will be in charge of this visit:

1. Maternal examination will comprise:

   * Inquiry of potential side effects (nausea, vomiting, diarrhea, rash, cough, peripheral edema, headache, abdominal pain, decrease appetite, others)
   * SAE/AE will be collected
   * Blood pressure measurement
   * Blood sampling: (5 ml) with: one Lithium Heparinate tube for letermovir dosage
   * 1 Heparinate Lithium tube (2 ml) for measurements of urea, creatinine, creatinine clearance, liver enzyme (ALAT ASAT GGT PAL), bilirubine
   * Hours of the 3 intakes of pills will be recorded in an individual treatment booklet
2. At TOP, fetal examination will comprise:

   * Fetal blood sampling (5 ml in a Lithium Heparinate tube for Letermovir dosage) collected at the time of feticide before lethal injection is given in the umbilical vein under ultrasound guidance.
   * Amniotic fluid sampling (5 ml on Lithium heparinate tube for Letermovir dosage) collected by the midwife at the time of artificial rupture of the amniotic membranes.
   * Placental biopsies sampling (2 cotyledons for Letermovir dosage) collected after delivery.
   * SAE/AE will be collected
3. At day 4 after TOP:

Phone call to collect SAE/AE after TOP

The duration of participation of each woman including data collection will be a maximum of 7 days (3 days before the TOP and 4 days after TOP).

The duration of the study will be 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman ≥ 18 years old
* in her second trimester of pregnancy
* undergoing TOP for any fetal abnormality
* no evidence of placental dysfunction.
* - affiliation to a social security regime//health insurance
* given consent for the study.
* patient must be able and willing to comply with study visits and procedures

Exclusion Criteria:

* Participation to another interventional drug trial (category 1)
* Subject protected by law under guardianship or curatorship
* Woman with creatinine clearance <75 ml/mn/1.73m2
* Woman with liver insufficiency (Child Pugh grade C), AST, ALT 5 x ULN, bilirubin 2 x ULN.
* Woman with known allergy to Letermovir
* Contraindication for the administration of Letermovir listed in the SmPC of Prevymis®
* Woman treated by pimozide, ergot alkaloids, dabigatran, atorvastatin, simvastatin, rosuvastatin, pitavastatine or cyclosporine.
* Concomitant administration of millepertuis
* Woman with hereditary intolerance to galactose, with lactose lapp deficiency, glucose or galactose malabsorption syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Concentrations reached in fetal blood relative to EC50 of letermovir. | At termination of pregnancy, on average 3 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Marianne LERUEZ-VILLE, PhD & MD, Study Chair — Virology laboratory- reference national Lab for CMV infection -Hôpital Necker-Enfants malades, Paris
Locations (1):
- Hôpital Necker - Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faure Bardon V, Peytavin G, Le MP, Guilleminot T, Elefant E, Stirnemann J, Leruez-Ville M, Ville Y. Placental transfer of Letermovir & Maribavir in the ex vivo human cotyledon perfusion model. New perspectives for in utero treatment of congenital cytomegalovirus infection. PLoS One. 2020 Apr 30;15(4):e0232140. doi: 10.1371/journal.pone.0232140. eCollection 2020. PMID 32353010